CLINICAL TRIAL: NCT06388356
Title: Patient's Informational Privacy in Prehospital Emergency Care: A Quasi-experimental Intervention Study
Brief Title: Patient's Informational Privacy in Prehospital Emergency Care - Educational Intervention Study for the Paramedics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eini Koskimies (Other)
Responsible Party: Sponsor-Investigator, Eini Koskimies, Doctoral reseacher, University of Turku
Organization: University of Turku (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 042024
Record Dates: First submitted 2024-04-19; First posted 2024-04-29 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Knowledge; Attitude of Health Personnel
Keywords: Informational privacy, confidentiality,

STUDY DESIGN:
Intervention Model Description: Two groups, intervention and control group. Only intervention group is receiveing the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Receives the educational intervention
  Interventions: Other: Educational intervention - Yksityisyyttä ensihoitoon / Informational privacy for preospital emergency care
- control group (No Intervention): The comparison group will not perform the educational intervention and will continue to work as normal standard according to their own organization's instructions.

INTERVENTIONS:
Other: Educational intervention - Yksityisyyttä ensihoitoon / Informational privacy for preospital emergency care — Educational intervention is a self-study, online course on Koulumaali platform about patient's informational privacy (IP) in prehospital emergency care (PEC).
  It comprises three separate educational modules approximately 30 min. long: module I) the meaning and significance of IP and its protection, module II) legislation regarding IP and its protection in healthcare and module III) breaches of IPand its protection in PEC.
  Each module contains theoretical sections as well as case-exercises and tests.
  Participants will have four weeks time to execute the entire course independently. Participants can execute the modules according to their own schedule. The modules need to be completed in certain order by following the numerical order from first to third. Only one of the modules is open at a time and the second module activates after the previous modules has been completed. Already completed modules become inactive.
  Arms: Intervention group

SUMMARY:
The main goal of this educational intervention study about patient's informational privacy (IP) is to evaluate the effect of the educational intervention into the paramedics' knowledge and attitude regarding patient's IP. The study also investigates the usability and the feasibility of the educational intervention.

The main questions it aims to answer are:

1. What is the effect of the educational intervention on the

   1. theoretical knowledge of paramedics' regarding IP?
   2. the paramedics' attitude towards patient's IP?
2. What is the usability and feasibility of the intervention being evaluated according to the respondents?

DETAILED DESCRIPTION:
The focus of this research is informational privacy (IP) in prehospital emergency care (PEC). The aim of this research is to improve the paramedics' knowledge of the patient's IP through an educational intervention. In addition, the educational intervention aims to impact positively to the paramedics' attitude towards patient's IP. The primary outcome of this research is the paramedics' knowledge about IP and the secondary outcome is the possible change in paramedics' attitude towards IP.

As a research method, a quasi-experimental research design with pre- and post-test with a comparison group is used. Sampling is purposive. Study is conducted in Finland. Advanced or basic support level paramedics working in two of the Finland's 21 rescue departments providing emergency medical services (EMS) in two of the wellbeing services counties in Finland is being recruited. These specific target rescue departments have been selected because of their similarity. Participants must also meet the separately defined inclusion criteria.

A simple random allocation is conducted to divide the rescue departments into intervention (n = 50 approximately) and control (n=50 approximately) group. Blinding is not conducted. Both, the researcher, and the participants will be aware about the result of the allocation.

The educational intervention is a self-study online course on Koulumaali (Moodle) platform about patient's IP in PEC. It includes three separate modules approximately 30 min. long: module I) the meaning and significance of IP and its protection, module II) legislation regarding IP and its protection in healthcare and module III) breaches of informational privacy and its protection in PEC. Each module contains theoretical sections as well as case-exercises and tests that allow participants to test their own skills.

The effectiveness of the educational intervention, the main and secondary outcomes, will be evaluated by the Knowledge and attitude towards patients' informational privacy (KAPIP) - instrument developed by the researcher, measuring the paramedics' subjective and actual (objective) theoretical knowledge about patient's IP as well as paramedics' attitude towards IP. In usability and feasibility evaluation, two separate questionnaires will be used. First, usability of the developed educational intervention will be measured by using the System Usability Scale (SUS), or more precisely its' Finnish version. The general feasibility of the educational intervention will be evaluated by using already existing questionnaire containing five structured items and three open ended questions. Permissions for the use of the already existing questionnaires has been received.

The research starts by recruiting the participants by email. An email is sent by separate contact persons from the target organizations to all the paramedics working in the target rescue departments in which they will be informed about the study, and how to take part in it if they meet the inclusion criteria presented in the information email. In addition, a privacy notice will be given. Possibility for further questions is also provided. In the information email targeted only for the participants in the intervention group, more precise description about performing the actual educational intervention is described.

Whether a paramedic is willing to participate to the study she/he will be asked to answer the electronic survey (KAPIP-instrument) to conduct the first measurement (pretest = M0). Link for the survey is provided in the information email. Informed consent and request for the email is placed at the beginning of the survey. Giving consent and email address is mandatory and controlled. Four weeks are set aside for the recruiting and the first measurement (pretest = M0).

The educational intervention will start right after the recruitment and first measurement. The intervention group will perform the educational intervention. The comparison group will not perform the educational intervention and will continue to work as normal standard according to the organization's instructions. Participants in the intervention group will receive instructions for completing the educational intervention from the contact person (researcher will inform the contact person regarding the participants to whom the instruction about the intervention execution needs to be sent). In total, the participants in the intervention group will have four weeks time to complete independently the educational intervention. Participants can execute the module according to their own schedule. The module does not have to be completed in one session and it can interrupt and resume the educational intervention later and continue at the same point. However, the modules need to be completed in certain order by following the numerical order from first to third. The educational intervention proceeds so that one of the modules is always open at a time. Participants' can evaluate their performance through tests and case exercises. The participant receives a mark of approval for the tests and case exercises performed automatically. If the respondent does not complete the modules, she/he will not be able to advance to the next module. Previously performed modules will be inactivated. This controls the correct and equal completion of the educational intervention. Researcher will monitor the participants' execution, and data regarding the execution times and how they perform the tasks will be collected from the Koulumaali platform (through Koulumaali activity monitoring). The last module of the educational intervention also includes the data collection regarding the participants' perceptions about the usability and feasibility of the educational intervention.

The second measurement (post-test = M1) phase starts right after the time (4 weeks) for the educational intervention execution has ended. Participants in control- and intervention group will receive an email from the target organizations' contact persons where they are asked to complete the same KAPIP-instrument within four weeks.

In the Evaluation phase of the intervention, the collected data is described and analysed. Apropriate statistical methods will be used; descriptive statistics (frequencies, proportions, mean, the standard deviation, meadians with lower and upper quantile) and statistical tests suitable for the data (linear mixed modes for repeated measures having group, time and group by time interaction in the model. In addition, cluster structure will be taken into account). Significance level of 0.05 (two-tailed) will be used and 95% confidence intervals will be calculated. Also, correlation analyses can be performed.

The research follows good scientific practice. An ethical approval is applied from The Ethics Committee for Health Care Division at the University of Turku and permissions for the study are applied from the target organizations.

Participants will be fully informed about the study and its phases in a separate information letters. In addition to the information letters, participants will be informed more precisely about the collection, processing, reporting and storing of data in the privacy statement form. All the collected data will be handled with appropriate manners and only by the research team including statisticians and possible research assistant. Only personal information necessary for the research will be collected. The personal data/sensitive information collected will be removed and coded with separate ID numbers before the data analysis (pseudonymization). Results will be reported in a way that it is not possible to identify individual respondents from the data. From the ethical point of view, it is also worth nothing, that the subjects are not representing particularly vulnerable group and they are taking part to the study voluntarily. Participation in research does not deviate from the principle of informed consent.

A separate data management plan has been conducted by using the DMPTuuli tool. In addition, a separate privacy notice informs respondents about the processing of their personal data. Both of these documents have been approved by The Ethics Committee for Health Care Division at the University of Turku.

ELIGIBILITY:
Inclusion Criteria:

* Participating paramedic has a degree in healthcare or is in the process of completing a health care degree.
* Participating paramedics is working as an ALS (advanced life support) or BLS (basic life support) level paramedic in one of the two target rescue departments during the entire time of the data collection.
* Participant is capable to understand Finnish.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-05-19 (Actual); Study Completion 2024-06-16 (Actual)

PRIMARY OUTCOMES:
Paramedics' knowledge about patient's informational privacy | Measurements are conducted during two different time frame: first measurement before the educational intervention taking up to 4 weeks. Second measurement after educational intervention taking up to 4 weeks.
  The possible change in paramedics' knowledge about patient's informational privacy (IP) will be evaluated by comparing the results from the first and second (after intervention) measurements from the both groups (experiment and control) by using the KAPIP (Knowledge and attitude towards patients' informational privacy) instrument developed for this research. It contains background factors and three separate sections. Sections I and II are providing the results for the main outcome:
  I) Subjective theoretical knowledge - paramedics' self-assessment of their knowledge about IP. Scaling from 1-5 (very poor, poor, fair, good, very good) II) Actual theoretical knowledge - knowledge test (objective evaluation regarding IP). Declarative sentences formed on true-or-false basis and with the option of I don't.
  The responses are scored as follows: In subjective and actual theoretical knowledge higher scores indicate higher level of knowledge: good, moderate, poor.

SECONDARY OUTCOMES:
paramedics' attitude towards patient's informational privacy. | Measurements are conducted during two different time frame: first measurement before the educational intervention taking up to 4 weeks. Second measurement after educational intervention taking up to 4 weeks.
  The possible change in paramedics' attitude towards patient's informational privacy will be evaluated by comparing the results from the first and second (after intervention) measurements from the both groups (experiment and control). The attitude will be assessed by using the KAPIP (Knowledge and attitude towards patients' informational privacy) instrument developed for this research. It contains background factors and three separate sections. Sections III is providing the results for the secondary outcome:
  III) Paramedics' attitude towards IP - 4-point Likert scale is used (1= Totally disagree 4 = totally agree).
  In the attitude section higher scores indicate more positive attitude.

CONTACTS AND LOCATIONS:
Overall Officials: Eini Koskimies, Doctoral researcher, Principal Investigator — University of Turku
Locations (1):
- University of Turku, Turku, Finland

REFERENCES:
- [Background] Brooke, J. (2013). SUS: A Retrospective. Journal of Usability Studies, 8(2), 29- 40. Brooke, J. (1996). SUS: a 'quick and dirty' usability scale. In: Usability evaluation in industry (Jordan PW, Thomas B, Weerdmeester BA, McClelland AL ed.), Taylor and Francis, London, pp. 189- 194.